CLINICAL TRIAL: NCT03696914
Title: Characteristics of the Eosinophilic Asthma Phenotype: an Observational Study in Patients From a Tertiary Care Center With Various Asthma Severities: The Quebec Heart and Lung Institute-Laval University Retrospective Asthma Database Analysis
Brief Title: Intense Airway Eosinophilia in Asthma
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Louis-Philippe Boulet, MD, FRCPC, Respirologist, Laval University
Other Study IDs: CÉR21488
Record Dates: First submitted 2018-10-02; First posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Asthma; Eosinophilic Asthma
Keywords: eosinophil; phenotype; cluster; asthma severity
MeSH Terms: conditions — Asthma; Pulmonary Eosinophilia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Eosinophilic: Asthmatic patients showing 3% or more sputum eosinophils
- Non-eosinophilic: Asthmatic patients showing less than 3% sputum eosinophils

SUMMARY:
In asthma, the type and importance of the inflammatory response in the airways has allows identification of different phenotypes. Of these, one of the most common is eosinophilic asthma, based on induced sputum differential cell count. Patients with severe asthma and an eosinophilic asthma phenotype have different pathophysiological characteristics than those seen in patients with with mild asthma. However, few studies have compared patients with eosinophilic phenotype according to the severity of asthma. In addition, the stability of the phenotype based on the sputum results has been criticized.

This study aims to describe the characteristics of patients with eosinophilic asthma phenotype according to the severity of asthma and determine the stability of the phenotype.

DETAILED DESCRIPTION:
Characteristics of asthmatic subjects with sputum eosinophilia will be compared according to asthma severity.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and over
* With a proven diagnosis of asthma as defined by one of the above criteria of current guidelines (36):

  1. Forced expiratory volume in one second (FEV1) increase by at least 12% (and ≥200 ml) after administration of a bronchodilator
  2. Current asthma symptoms and a methacholine provocative concentration inducing a 20% fall in FEV1 (PC20) <16 mg/ml
  3. A respirologist's current diagnosis of asthma found in the patient's medical report 3. Non-smokers or smokers/ex-smokers defined as someone with a smoking history <10 pack-years 4. With sputum differential cell count result 5. Considered to receive optimal treatment for their disease (as per current guidelines except for patients included in exploratory objective 1.

     6. Stable asthma and asthma medication for at least 4 weeks before data analysis 7. Written informed consent obtained for inclusion in the database

     Exclusion Criteria:
     1. Any respiratory disease apart from asthma
     2. Current or ex-smokers should not have a smoking history ≥10 pack-year before data analysis. Patients who administer nicotine in other forms (patches, chew tobacco, e-cigarette, etc.) will be excluded
     3. Unstable asthma medication <4 weeks before data analysis
     4. Asthma exacerbation (see definition below) <4 weeks before data analysis
     5. Respiratory tract infection <4 weeks before data analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthmatic subjects from the Quebec city region.
Sampling Method: Non-Probability Sample
Enrollment: 918 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-08-03 (Actual)

PRIMARY OUTCOMES:
Asthma severity according to medication use | Baseline
  Prevalence of patients with 3% or more sputum eosinophils in mild, moderate and severe asthma

SECONDARY OUTCOMES:
ACSS symptom sub-score | Baseline
  Comparison of asthma control between patients with 3% or more sputum eosinophils and patients with less than 3% sputum eosinophils
FEV1 percent predicted | Baseline
  Comparison of forced expiratory volume in one second between patients with 3% or more sputum eosinophils and patients with less than 3% sputum eosinophils

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Philippe Boulet, MD, Principal Investigator — IUCPQ-UL
Locations (1):
- Centre de recherche de l'Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No